CLINICAL TRIAL: NCT03769714
Title: A Placebo-controlled, Double-blinded, Randomized Pilot Study of Bupivacaine Liposome Injectable Suspension (EXPAREL) for Minimally Invasive Supracervical Hysterectomies Postsurgical Analgesia
Brief Title: EXPAREL for Minimally Invasive Supracervical Hysterectomies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-02-12-MMC
Record Dates: First submitted 2018-08-22; First posted 2018-12-07 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Pain
Keywords: laparoscopy; supracervical hysterectomy; Multimodal pain management; bupivacaine liposome; Exparel
MeSH Terms: conditions — Pain | interventions — Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline Solution for Injection (Active Comparator): Group A (control, n=26) to receive 20ml of saline while prepping. The syringe will covered as to disguise the contents of the syringe.
  Interventions: Drug: Saline Solution for Injection
- Exparel (Experimental): Group B (study, n=26) to receive 20ml of liposomal bupivacaine (EXPAREL) into the stroma of the cervix at the 4 and 8 o'clock positions (innervation insertion points of the cervix).
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Saline Solution for Injection — Injection of 20mL of 0.9%Normal Saline
  Other Names: Standard
  Arms: Saline Solution for Injection
Drug: Exparel — Exparel (bupivacaine liposome injectable suspension) is a liposome injection of bupivacaine, an amide-type local anesthetic, indicated (bupivacaine liposome injectable suspension) for administration into the surgical site to produce postsurgical analgesia.
  Other Names: liposomal bupivicaine
  Arms: Exparel

SUMMARY:
The aim of the of the study is a reduction in minimally invasive supracervical hysterectomy postsurgical pain, which may result in less need for supplemental opioid pain medications, fewer opioid related adverse events, and a better recovery experience for patients, which may offer an economic benefit to health care systems.

Intracervical preoperative dose of Exparel during minimally invasive (robotic--assisted or traditional laparoscopy) supracervical hysterectomy reduces cumulative pain scores for up to 24 hours and reduces overall requests for break through (additional) analgesia with opioid consumption compared with placebo.

DETAILED DESCRIPTION:
Exparel is a local analgesic that utilizes bupivacaine in combination with the proven product delivery platform, DepoFoam®. Exparel (bupivacaine liposome injectable suspension) is a liposome injection of bupivacaine, an amide-type local anesthetic, indicated (bupivacaine liposome injectable suspension) for administration into the surgical site to produce postsurgical analgesia. Liposomal drug- containing formulations can provide for controlled drug release over an extended period of time.

The overall length of hospital stay (LOS) for patients undergoing laparoscopic (robot- assisted or traditional laparoscopy) supracervical hysterectomy varies widely in published reports; typical durations range between 0 days and 4 days.

That is because in recent years there has been a trend toward use of enhanced or "fast- track" discharge protocols to reduce LOS in patients undergoing this procedure, predicated primarily on reducing the time to achieve tolerance of oral liquid/food intake and improved GI function. Most patients experience moderate to extreme pain after surgery and effective postsurgical pain management is a key factor affecting patient recovery. Multimodal analgesia techniques involving analgesics, such as local anesthetics, oral or parenteral nonsteroidal anti-inflammatory medications, and oral or parenteral opioids, are recommended as the safest and effective approach to postsurgical pain control. Local anesthetics administered during surgery are frequently used as part of multimodal analgesic regimens; however, the duration of analgesia with these agents is short (12 hours). Bupivacaine has a long history of use in the surgical setting, and the efficacy of bupivacaine HCl administered perioperatively via wound infiltration or acute postsurgical pain is well established. A novel formulation of bupivacaine, ie, liposome bupivacaine (Pacira Pharmaceuticals, Inc., Parsippany, NJ), has been developed to address the need for longer-acting local anesthetics that can be administered as a single dose. The question becomes whether this drug is effective for postsurgical analgesia if given preoperatively via the intracervical stroma during minimally invasive gynecologic surgical procedures, specifically laparoscopic (robot--assisted or traditional laparoscopy) supracervical hysterectomy.

Paracervical/intracervical injections are used for cervical/uterine manipulation in various obstetrical and gynecological procedures. Lukas et al used the intracervical/paracervical block prior to hysteroscopic polypectomy, with good pain scores following the procedure and no serious adverse effects were noted. In addition, Chauan et al also noted good pain control with intracervical injection with lidocaine in patients undergoing a hysterosalpingography, which involves distended the uterus and injecting dye. Mankowshi et al also studied both intracervical and paracervical injections of lidocaine for first trimester suction curettage and found no difference between the two forms ensuring that both effective means of analgesia.

In the U.S., surgical site infections (SSI) affect 1 in 24 patients that undergo inpatient surgery. Most surgical site infection take place after day 5 , which will be out of the scope of timeframe for conduct of the survey. However a SSI can make the differentiation of pain from the surgery itself and pain from a complication of surgery difficulty to differentiate. The patient will be asked to specify where the pain is and ask if they have any associated vaginal discharge, foul smelling odor, and difficulty urinating and or passing a bowel movement. These responses will be tracked, and if the participant shows signs of a SSI, the patients may warrant a closer followup in the office and or asked to go directly to the Emergency Department (ED). The patients will still be included in the study but special note will be made of how many participant had SSI in the discussion portion.

Methods:

Randomized double blind placebo controlled pilot study. After IRB approval, 52 subjects will be consented to participate in the study. The study includes subjects undergoing minimally invasive (robot--assisted or traditional laparoscopy) supracervical hysterectomy under general anesthesia. This study will include women (35 - 75 years) who have American Congress of Obstetricians and Gynecologists (ACOG) and American Association of Gynecologic Laparoscopists (AAGL) physical classification status for a minimally invasive (robotic- assisted or traditional laparoscopy)supracervical hysterectomy.

Randomization will be done prior to recruitment of patient via computer software. There will be two groups with numbers 1-52, no numbers will be repeated. Each patient that is recruited will be assigned a number from 1-52 (in sequential order); the master list will be kept with the pharmacy director. Group A (control, n=26) to receive 20ml of saline while Group B (study, n=26) to receive 20ml of liposomal bupivacaine (EXPAREL) into the stroma of the cervix at the 4 and 8 o'clock positions (innervation insertion points of the cervix).

The MMC Pharmacy will prepare an individualized numbered bubble wrapped amber package accordingly to the randomization. It will be prepared prior to the recruitment and kept in the fridge in 4th floor PACU pharmacy. After the patient is consented and given a subject number, the package with the corresponding number will be picked up from the pharmacy and given to either the resident/attending (not involved in the study) who will share the contents of the package with the anesthesia team. While prepping, the same individual will inject the contents. The syringe will covered as to disguise the contents of the syringe.

The investigators will show a short video on how to prepare the Exparel as well the injection component in order to diminish the differences between the individuals.

Measurements:

The severity of pain will be assessed preoperatively in the holding area, PACU arrival, 12, 24, and 48 hours postoperatively using a numeric rating scale (NRS) at rest for pain with 0 = no pain and 10 = worst possible pain. Pain inquiries will assess low pelvic/suprapubic area and lower abdominal pain, type of pain (dull, achy, sharp, stabbing, etc.) and radiation of pain to a surrounding area. Other endpoints will include number of patients who required break through (additional) opioid analgesic medications, median time to first break through opioid use, total opioid analgesic requirement. The time, day and number of requests for break through (additional) analgesia will be noted by gynecologic surgery team (Resident or Fellow) participating in this study.

When the patient is home the patient will have a Pain Medication Diary that the investigators will provide for the patient prior to discharge. The patient will bring at the post-operative visit and or mail it in.

ELIGIBILITY:
Inclusion Criteria:

1. 35--75 years of age at the Screening Visit.
2. Female subjects only.
3. Scheduled to undergo minimally invasive (robotic-assisted or laparoscopic) supracervical hysterectomy, under general anesthesia.
4. Clinical laboratory values less than twice the upper limit of normal or, if abnormal, deemed not clinically significant per the Investigator.
5. Ability to provide informed consent, adhere to the study visit schedule and complete all study assessments and language specific questionnaires.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant.
2. Use of any of the following medications within the times specified before surgery: a. opioid, SSRI, tricyclic antidepressant, gabapentin, pregabalin within three days of surgery. b. Use of acetaminophen within 24 hours of surgery.
3. Concurrent painful physical condition or concurrent surgery that may require analgesic treatment (such as NSAID, opioid, SSRI, tricyclic antidepressant, gabapentin, pregabalin) in the postoperative period for pain that is not strictly related to the minimally invasive supracervical hysterectomy procedure and may confound the postoperative assessments (e.g., rheumatoid arthritis, chronic neuropathic pain.
4. Chronic user of analgesic medications, including taking opioid medications for more than 14 days in the last 3 months, or non-opioid pain medications more than 5 times per week.
5. Current use of systemic glucocorticosteroids (e.g. Decadron) or use of glucocorticoids within one month of enrollment into this study.
6. History of hepatitis (other than hepatitis A).
7. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
8. Failure of presurgical drug and alcohol screen.
9. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics, opioids, or propofol.
10. Administration of an investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

12. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance. 13. Significant medical conditions or laboratory results that, in the opinion of the Investigator indicate an increased vulnerability to study drug and procedures, and expose subjects to an unreasonable risk as a result of participating in this clinical trial. 14. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postoperative course. 15. An incision length greater than 3 cm.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Bral, M.D., Principal Investigator — Minimally Invasive Surgery -Fellowship Director
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Result] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Result] White PF. Multimodal analgesia: its role in preventing postoperative pain. Curr Opin Investig Drugs. 2008 Jan;9(1):76-82. PMID 18183534
- [Result] Smoot JD, Bergese SD, Onel E, Williams HT, Hedden W. The efficacy and safety of DepoFoam bupivacaine in patients undergoing bilateral, cosmetic, submuscular augmentation mammaplasty: a randomized, double-blind, active-control study. Aesthet Surg J. 2012 Jan;32(1):69-76. doi: 10.1177/1090820X11430831. Epub 2011 Dec 16. PMID 22179931
- [Result] Portillo J, Kamar N, Melibary S, Quevedo E, Bergese S. Safety of liposome extended-release bupivacaine for postoperative pain control. Front Pharmacol. 2014 Apr 30;5:90. doi: 10.3389/fphar.2014.00090. eCollection 2014. PMID 24817851
- [Result] Chudnoff S, Einstein M, Levie M. Paracervical block efficacy in office hysteroscopic sterilization: a randomized controlled trial. Obstet Gynecol. 2010 Jan;115(1):26-34. doi: 10.1097/AOG.0b013e3181c51ace. PMID 20027030
- [Result] Lukes AS, Roy KH, Presthus JB, Diamond MP, Berman JM, Konsker KA. Randomized comparative trial of cervical block protocols for pain management during hysteroscopic removal of polyps and myomas. Int J Womens Health. 2015 Oct 13;7:833-9. doi: 10.2147/IJWH.S50101. eCollection 2015. PMID 26543383

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Solution for Injection: Group A (control, n=30) to receive 20ml of saline while prepping. The syringe will covered as to disguise the contents of the syringe.
  Saline Solution for Injection: Injection of 20mL of 0.9%Normal Saline
- Exparel: Group B (study, n=30) to receive 20ml of liposomal bupivacaine (EXPAREL) into the stroma of the cervix at the 4 and 8 o'clock positions (innervation insertion points of the cervix).
  Exparel: Exparel (bupivacaine liposome injectable suspension) is a liposome injection of bupivacaine, an amide-type local anesthetic, indicated (bupivacaine liposome injectable suspension) for administration into the surgical site to produce postsurgical analgesia.
Period: Overall Study
Arm/Group | Saline Solution for Injection | Exparel
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Solution for Injection | Exparel | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 47 [44 to 50] | 45 [43 to 49] | 46 [43 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Pain at 12 Hours
Description: Participant will be shown a card that has a visual analogue (Faces) pains scale combined with numerical (0-10) analogue scale (0 is no pain, 10 is the worst pain imaginable).at 12 hours postoperatively
Time Frame: 12 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Solution for Injection | Exparel
Number analyzed (Participants) | 27 | 28
score on a scale | 3.9 (3.1) | 3.7 (2.9)

2. Primary Outcome: Pain at 48 Hours
Description: Participant will be shown a card that has a visual analogue (Faces) pains scale combined with numerical (0-10) analogue scale (0 is no pain, 10 is the worst pain imaginable).at 48 hours postoperatively
Time Frame: 48 hours after surgey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Solution for Injection | Exparel
Number analyzed (Participants) | 24 | 26
score on a scale | 3.2 (2.2) | 3.9 (1.8)

ADVERSE EVENTS:
Time Frame: 48 hours
Description: adverse events
Arm/Group | Saline Solution for Injection | Exparel
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03769714/Prot_000.pdf